CLINICAL TRIAL: NCT01995331
Title: Moderate-dose Cyclophosphamide for Childhood Acquired Aplastic Anemia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Xiaofan Zhu (Unknown)
Responsible Party: Sponsor-Investigator, Xiaofan Zhu, chief physician, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YL20102601
Record Dates: First submitted 2013-11-21; First posted 2013-11-26 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-11

CONDITIONS: Aplastic Anemia
Keywords: aplastic anemia;; cyclophosphamide;; immunosuppressive therapy;; cyclosporine A
MeSH Terms: conditions — Anemia, Aplastic | interventions — Cyclophosphamide; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- moderate-dose cyclophosphomide (Other)
  Interventions: Drug: cyclophosphamide,cyclosporine A

INTERVENTIONS:
Drug: cyclophosphamide,cyclosporine A — Drug,cyclophosphamide,cyclophosphamide (30 mg/kg/day) administered intravenously (IV) over 1 hr for 4 consecutive days Drug,cyclosporine A,5mg-12mg/kg.d,CSA was administered orally 40 days after the fourth dose of cyclophosphamide and maintained for 3 years. The dose of CSA was adjusted to maintain trough drug concentration above 150 μg/L and peak drug concentration above 300 μg/L.
  Drug, human granulocyte colony-stimulating factor (rhG-CSF), 5 μg/kg/day subcutaneously starting 24 hrs after the fourth dose of cyclophosphamide, and it was withdrawed when ANC was >1×109/L.
  Other Names: Drug,Mesnaum

SUMMARY:
Severe aplastic anemia (SAA)is characterized by the depletion of hematopoietic precursors associated with life-threatening complications. High-dose cyclophosphamide has been found to yield a complete response (CR) in adults and children with SAA.However, the optimal dosage of cyclophosphamide for patients in childhood remains unclear. So we explore the ideal dosage of cyclophosphamide for the treatment of children with SAA.

DETAILED DESCRIPTION:
Tisdale et al. (2000,2002) attempted to compare immunosuppression using ATG/CSA with high-dose cyclophosphamide (50 mg/kg/d for 4 consecutive days) plus CSA in a randomized trial of newly diagnosed adults with SAA. Both groups received CSA as part of the treatment regimen. However, the trial was terminated prematurely due to excessive morbidity among the patients treated in the cyclophosphamide arm. They documented that invasive fungal infections were severe among the cyclophosphamide group. Between January 2008 through May 2009, in our department, nine pediatric patients with a diagnosis of SAA were enrolled a study with lower dose of cyclophosphamide with 30mg/kg/day for 4 consecutive days and combination with CSA, this study shows promise for children with severe aplastic anemia.Now we want explore the dosage of cyclophosphamide.

ELIGIBILITY:
Inclusion Criteria:

* Acquired Childhood Severe Aplastic Anemia (SAA)

Exclusion Criteria:

* not Childhood and Acquired Severe Aplastic Anemia

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-03; Primary Completion 2015-03 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
The reponse of Moderate-dose Cyclophosphamide for Childhood Acquired Aplastic Anemia | 36 months
  Complete response (CR) was defined as achieving normal levels of hemoglobin adjusted for age, platelet count >100×109/L, and ANC>1.5×109/L. Partial response (PR) was defined as transfusion independence, reticulocyte count >30×109/L, platelet count >30×109/L, and ANC >0.5×109/L above the baseline. Persistence of transfusion requirement or death was evidence of no response (NR).

SECONDARY OUTCOMES:
The side effect of Moderate-dose Cyclophosphamide for Childhood Acquired Aplastic Anemia | 36 months
  To report the death rate and the death cause , the infection rate and the pathogenic bacteria, especialy the fungal infection rate.
  To report other toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaifan Zhu, MD, Principal Investigator — Department of Pediatrics, Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Department of Pediatrics,Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Tianjin, Tianjin Municipality, China